CLINICAL TRIAL: NCT04820751
Title: Cyproheptadine in Severe COVID-19 : A Unblinded Randomized Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Covid-19 Early Treatment Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25584
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Viral Pneumonia; Serotonin Syndrome; Platelet Dysfunction
Keywords: Covid 19
MeSH Terms: conditions — Pneumonia, Viral; Serotonin Syndrome; COVID-19 | interventions — Cyproheptadine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyproheptadine and standard care (Experimental): Start Cyproheptadine 8mg three times a day during 5 days. Dose will be reduced to 4mg three times a day if GFR inferior to 30ml/min/1.73m²
  Standard management of COVID-19 infection according to current international guidelines
  Interventions: Drug: Cyproheptadine Hydrochloride 4 MG
- Standard care (No Intervention): Standard management of COVID-19 infection according to current international guidelines

INTERVENTIONS:
Drug: Cyproheptadine Hydrochloride 4 MG — Cyproheptadine associated to standard care
  Other Names: Standard Care
  Arms: Cyproheptadine and standard care

SUMMARY:
This randomized controled open label clinical trial is to evaluate the effect of Cyproheptadine on the clinical course of patients presenting a severe SARS-COV 2 pneumonia.

DETAILED DESCRIPTION:
Observational and biochemical studies have identified an interesting pathway in the pathophysiology of certain clinical-biological characteristics of COVID-19, linked to an excess of serotonin. We hypothesize that the antagonism of the action of serotonin could improve the clinical course of patients most severely affected by COVID-19.

One such antagonist of serotonin with a long track record of safety and tolerability is cyproheptadine. Cyproheptadine acts as an antagonist of 5-hydroxytryptamine (5HT=serotonin) receptor subtype 2 as well as histamine-1 receptor. Many of the potent effects of serotonin on lung vascular tone, respiratory rate, and systemic vascular beds are mediated by 5-HT receptor subtype 2.

Investigators will randomize approximately 200 participants, aged 18 and older, who have tested positive for COVID-19 and who will be hospitalized at Santa Cabrini Hospital in Montreal, Quebec, Canada, presenting a severe form of covid-pneumonia-19 requiring supplemental oxygen.

Study eligibility of all participants will be assessed first. Once a participant is confirmed eligible and consented, they will participate in the study.

Participants will be randomly assigned (1: 1) to either take cyproheptadine 8 mg by mouth three times a day for 5 days and receive standard care or receive standard care alone.

The dose will be adjusted according to the glomerular filtration rate.

On D1, D3, D5, D7 and D10 since randomization, participant's vital signs (including SpO2, respiratory rate, FiO2 or oxygen flow, heart rate, blood pressure and temperature), blood creatinine, bilirubin, CRP, LDH, Dimers and platelets the count will be evaluated. Any adverse event will be assessed daily and documented.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 or older
* Hospitalized and requiring medical care for COVID-19
* Presenting respiratory failure cause by COVID 19 requiring oxygen and/or mechanical ventilation support
* With radiographic evidence of pulmonary infiltrate
* Able to give informed consent or, if unable to do so regarding the medical condition, having relatives able of consenting for the patient

Exclusion Criteria:

* Pregnancy
* Patients with pre-existing terminal condition with life expectancy < 6 months
* Patients with pre-existing severe lung disease requiring home O2
* History of seizure disorder
* History of adverse reaction to antihistamines or to Cyproheptadine

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-10 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Length of hospitalization | Through study completion, an average of 1 year
Need mechanical ventilation (Non invasive or Invasive) | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Death | Day 28
Length of hospitalization in the intensive care unit | Through study completion, an average of 1 year
Duration of mechanical ventilation | Through study completion, an average of 1 year
SOFA Score | At Day 1,3,5,7,10 after randomization
  Sequential Organ Failure Min Score 0-Max score 24 Higher scores mean a worse outcome
Heart rate | At Day 1,3,5,7,10 after randomization
Respiratory Rate | At Day 1,3,5,7,10 after randomization
Spo2/FiO2 and ROX ratio | At Day 1,3,5,7,10 after randomization
CRP level | At Day 1,3,5,7,10 after randomization
LDH level | At Day 1,3,5,7,10 after randomization
D-Dimere level | At Day 1,3,5,7,10 after randomization
Platelet count | At Day 1,3,5,7,10 after randomization